## Statistical Plan

## 1. Baseline data

Descriptive data on sample demographics, injury characteristics (e.g., GOS-E), and symptom and process measures (ESS, FSS, FOSQ, SEMSA, OTBQ) will be presented at M(SD) for continuous data and count (%) for categorical data.

## 2. Outcome Measures

Quantitative study outcome measures (e.g., ESS, FSS, FOSQ) will be presented at M(SD) for continuous data. Qualitative data (NEII) will be analyzed using thematic analysis and a constant comparative approach, with two team members independently reviewing transcripts and applying codes. Summary of recruitment, retention, and missingness on measures will be presented. Distributions of  $\leq \pm 2.0$  for skewness and  $\leq \pm 7.0$  for kurtosis will be considered sufficiently normal. Effect sizes for change scores on symptom measures will be measured using Cohen's d with correction for small sample sizes with 95% confidence intervals